CLINICAL TRIAL: NCT05603390
Title: Heart Failure With Mildly Reduced Ejection Fraction Registry (HARMER)
Brief Title: Heart Failure With Mildly Reduced Ejection Fraction Registry
Acronym: HARMER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Michael Behnes, Prof. Dr. med. Michael Behnes, Universitätsmedizin Mannheim
Other Study IDs: 2022-818
Record Dates: First submitted 2022-10-10; First posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Heart failure (HF) affects about 1% of patients younger than 55 years, whereas the prevalence of HF increases > 10% in patients with at least 70 years of age. Despite HF with reduced ejection fraction (HFrEF) and HF with preserved ejection fraction (HFpEF), the clinical significance of HF with mildly reduced ejection fraction (HFmrEF) has gained more importance within the past years. Those patients are characterized by a left ventricular ejection fraction (LVEF) of 41-49%. However, within the current European guidelines, limited treatment recommendations in this subgroup of HF are yet available as a consequence of the limited number of studies in this field. The "Heart Failure With Mildly Reduced Ejection Fraction Registry" aims to characterize patients with HFmrEF and investigated the prognostic impact of interventional and pharmacological therapies in this subgroup of HF patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HFmrEF (i.e., LVEF 41-49%)
* Patients with at least 18 years of age

Exclusion Criteria:

* Patients younger than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The present study consecutively includes patients with heart failure with mildly reduced ejection fraction (HFmrEF) from 2015 to 2022.
Sampling Method: Probability Sample
Enrollment: 2200 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 2 years.
  All-cause mortality

SECONDARY OUTCOMES:
Change of LVEF | 2 years.
  Change of LVEF
Change of NT-pro BNP | 2 years.
  Change of NT-pro BNP
Heart-failure related hospitalization | 2 years.
  Heart-failure related hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Michael Behnes, MD, Principal Investigator — First Department of Medicine, University Medical Centre Mannheim, Germany.
Locations (1):
- University Medical Centre Mannheim, Mannheim, Germany

REFERENCES:
- [Derived] Schmitt A, Akin I, Reinhardt M, Abel N, Lau F, Dudda J, Abumayyaleh M, Weidner K, Bertsch T, Duerschmied D, Behnes M, Schupp T. Albumin, urea-to-albumin ratio, or the albumin-to-creatinine ratio to predict outcomes in heart failure with mildly reduced ejection fraction. Eur J Clin Invest. 2026 Jan;56(1):e70165. doi: 10.1111/eci.70165. Epub 2025 Dec 26. PMID 41452958
- [Derived] Reinhardt M, Behnes M, Weidner K, Abumayyaleh M, Lau F, Schmitt A, Abel N, Duerschmied D, Weiss C, Akin M, Akin I, Schupp T. Prognostic Implications of Sex in Patients With Heart Failure With Mildly Reduced Ejection Fraction: Results From a Large-Scaled Registry. J Am Heart Assoc. 2025 Jan 21;14(2):e033173. doi: 10.1161/JAHA.123.033173. Epub 2025 Jan 16. PMID 39817535